CLINICAL TRIAL: NCT06215768
Title: Comparative Study of Preoperative Intravenous Dexmedetomidine Versus Preoperative Intravenous Midazolam On the Incidence of Emergency Delirium in Pediatric Patients Undergoing Tonsillictomy and Adenoidectomy a Prospective Randomized Clincal Trial
Brief Title: Emergency Delirium in Pediatrics Undergoing Tonsillectomy and Adenoidectomy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Esraa Abdel Azez Soltan Mohamed Zayed (Other)
Responsible Party: Sponsor-Investigator, Esraa Abdel Azez Soltan Mohamed Zayed, Director, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Emergency delirium
Record Dates: First submitted 2024-01-06; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Emergence Delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexemedetomidine group A (Experimental): Patients aged( 2_12) years, American Society of Anesthesiologists class (ASA) I or II, scheduled for tonsillectomy with and without adenoidectomy will be randomized to receive intravenous dexmedetomidine 0.5 μg/kg
  Interventions: Drug: Dexmedetomidine and Midazolam
- Midazolam group B (Experimental): Patients aged( 2_12) years, American Society of Anesthesiologists class (ASA) I or II, scheduled for tonsillectomy with and without adenoidectomy will be randomized to receive intravenous midazolam 0.1 mg/kg
  Interventions: Drug: Dexmedetomidine and Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine and Midazolam — This will be a prospective, double-blind, randomized controlled study conducted between October 2023and June 2024 .
  Patients aged( 2_12) years, American Society of Anesthesiologists class (ASA) I or II, scheduled for tonsillectomy with and without adenoidectomy will be randomized to receive intravenous dexmedetomidine 0.5 μg/kg Or intravenous midazolam 0.1 mg /kg(Group A) or (Group B) over 10 minutes after induction of anesthesia. The primary outcome is the incidence of ED within 30 minutes after extubation. Other outcomes are the incidence of pain, extubation time, post-anesthesia care unit (PACU) length of stay after extubation, adverse events, and the incidence of negative postoperative behavioral changes (NPOBCs).

SUMMARY:
Primary outcom Compare the effectiveness of study drugs on reducing the incidence of emergence delirium .

Secondary outcomes:

Sedation score Intensity of pain by FLACC Extubation time Iength of stay in Post anesthetic care unite (PACU ) Incidence of negative post operative behavioural changes (NPOBCs ) Laryngeospasm ny adverse effects

DETAILED DESCRIPTION:
Emergence delirium (ED) is a common neurologic complication that can not only distress children and their families in the early postanesthetic period, but can also have adverse effects on children in the long-term Emergence delirium (ED) is an acute confusion state during recovery from anesthesia; patients with ED may present with disorientation, hallucination, restlessness, and purposeless hyperactive physical behavior . ED is not fully equivalent to EA; ED can involve hypoactive signs or mixed forms and hyperactive signs similar to agitation . Nevertheless, the terms EA and ED have been used interchangeably in several studies Pediatric patients undergoing tonsillectomy and adenoidectomy usually have a high incidence of POED, which increases the risk of developing postoperative airway obstruction and respiratory depression due to anatomical characteristics of operative location and increased susceptibility to opioid analgesics.

Postoperative emergence delirium develops in 12% to 18% of all children undergoing general anesthesia for surgery.

dexmedetomidine, is a selective alpha-2 agonist, which works in the brain and spinal cord that has sedative, analgesic and anxiolytic properties. Dexmedetomidine also has the ability to lower the overall anesthetic requirements by reducing sympathetic outflow in response to painful surgical stimulation.

Midazolam is a widely used intravenous anesthetic agent with rapid onset, short duration of action and relatively rapid plasma clearance. It is mainly used to produce preoperative sedation and the induction of general anesthesia The action of midazolam can be explained through its action on gammaaminobutyric acid (GABA) receptors. GABA receptors mediate inhibitory neurotransmission in the central nervous system In our study we aim to compares the effectiveness of preoperative intravenous dexmedetomidine versus intravenous midazolam for the prevention of emergence delirium in pediatric patients undergoing tonsillectomy , adenoidectomy or both . .

ELIGIBILITY:
Inclusion Criteria:

- Pediatric patients aged 2-12 years

With ASA physical status 1 or 2

Who were scheduled for tonsillectomy with and without adenoidectomy under general anesthesia

Exclusion Criteria:

* Emergency surgery

Intellectual disability

Neurological disease

Renal , hepatic, cardiac or respiratory disease

Allergy to the study drugs

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Emergency Delirium | 30 minutes
  The incidence of emergence delirium in pediatrics undergoing tonsillectomy and adenoidectomy a prospective randomised clinical trial .

SECONDARY OUTCOMES:
FLACC | 30 minutes
  Measure of intensity of pain by face , legs ,activity Cry , consolability

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Hassanen, Study Director — Department of anesthesia , intensive care and pain management